CLINICAL TRIAL: NCT04404049
Title: The HIV Functional Cure Potential of UB-421: A Phase II, Randomized, Open-label, Controlled, 48 Week, Proof of Concept Study, to Evaluate the Safety of UB-421 in Combination With Standard Antiretroviral Therapy (ART) and the Efficacy of HIV Reservoir Reduction as Compared With ART Alone in ART Stabilized HIV-1 Patients
Brief Title: The HIV Functional Cure Potential of UB-421 in ART Stabilized HIV-1 Patients
Acronym: HIV-1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: UBP Greater China (Shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UBP-A218-HIV
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — UB-421

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard ART (No Intervention): Subjects will receive standard ART for 48 weeks
- UB-421(25mg/kg) Q2W add-on treatment (Experimental): UB-421(25 mg/kg) Q2W plus standard ART for 48 weeks
  Interventions: Biological: UB-421(25 mg/kg) Q2W
- UB-421(25mg/kg) Q4W add-on treatment (Experimental): UB-421(25 mg/kg) Q4W plus standard ART for 48 weeks
  Interventions: Biological: UB-421(25 mg/kg) Q4W

INTERVENTIONS:
Biological: UB-421(25 mg/kg) Q2W — Monoclonal antibody by IV infusion plus standard ART
  Arms: UB-421(25mg/kg) Q2W add-on treatment
Biological: UB-421(25 mg/kg) Q4W — Monoclonal antibody by IV infusion plus standard ART
  Arms: UB-421(25mg/kg) Q4W add-on treatment

SUMMARY:
This is a Phase II, randomized, open-label, multi-center, active-controlled study to assess the safety, tolerability, and efficacy of UB-421 administered as an add-on to the standard ART in ART-treated HIV-1 subjects with stably suppressed HIV-1 plasma VL. The study will be conducted at multiple study centers, designated AIDS hospitals in China.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 sero-positive
2. Male with body weight ≥ 50 kg or female with body weight ≥ 45 kg.
3. HIV-1 plasma RNA level below 50 RNA copies/mL.

Exclusion Criteria:

1. Subjects with active systemic infections, except for HIV-1, that the Investigator feels the infections may confound evaluation and treatment for HIV-1.
2. Current active hepatitis B carriers, ie, hepatitis B surface antigen positive.
3. Current active hepatitis C carriers, ie, hepatitis C virus (HCV) antibody positive.
4. History of anaphylaxis to other mAbs.
5. Any vaccination within 8 weeks prior to the first dose of assigned drug.
6. Use of immunomodulators, HIV vaccine, or systemic chemotherapy within 180 days prior to the first dose of assigned drug.
7. Females who are pregnant, lactating, or breastfeeding, or who plan to become pregnant during the study.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
treatment related TEAEs | 48Weeks
  the incidence of Grade 3 drug-related treatment-emergent adverse events

SECONDARY OUTCOMES:
the change of immune profiles | 16Weeks
  Change in Treg percentage in the peripheral blood